CLINICAL TRIAL: NCT03818438
Title: Biomechanical Analysis, Complementary Examinations and Rehabilitative Management of Chronic Ankle Instability
Brief Title: Chronic Ankle Instability Diagnostic Tests Determining Underlying Deficits
Acronym: CAIDiag
Status: Terminated | Type: Observational
Why Stopped: insufficiency inclusion; covid crisis ; sponsor decision
Sponsor: University Hospital, Lille (Other)
Collaborators: Ministry of Health, France (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2017_09; 2018-A00102-53 (Other: ID-RCB number, ANSM)
Record Dates: First submitted 2019-01-09; First posted 2019-01-28 (Actual); Last update posted 2022-05-31 (Actual); Status verified 2022-05

CONDITIONS: Ankle Dislocation; Chronic Ankle Instability
Keywords: Chronic instability; Strength; Proprioception; Rehabilitation; Ankle; Balance

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Case subjects adult patients with chronic ankle instability: Male or female subjects aged 18-45, presenting :
  * at least one acute lateral ankle sprain (i.e. initial ankle sprain more than 12 months before inclusion),
  * at least one residual symptom (giving way OR sensation of instability OR recurrent ankle sprain), confirmed by a score < 24 on the Chronic Ankle Instability Tool (CAIT)
  * Impact on activities of daily living and sport, score < 90% on Foot and Ankle Ability Measure (FAAM) and < 80% on FAAM-sport Case subjects are free of any other lower extremity pathologies or pain Subjects presenting bilateral chronic ankle instability are excluded
- Healthy subjects: Male or female subjects aged 18-45 (matched with case Healthy subjects), without any lower extremity pathologies

SUMMARY:
Chronic ankle instability is a common condition in the active adult population and characterized by the occurrence of repeated giving way and/or recurrent ankle sprains. Multiple underlying deficits have been proposed, among which ankle muscle strength deficits, proprioception deficits, ( static and dynamic balance disorders, and articular laxity. Unfortunately, no consensus exists on which clinical tests should be realized to determine if one of these underlying deficits is predominant and as a result could guide the rehabilitation process. The study hypothesis is that people with chronic ankle instability might be heterogenous and could be divided in different subgroups as a function of underlying deficits. Therefore, this study aims to evaluate the capacity of different clinical tests to differentiate people with chronic ankle instability from healthy people as well as between each other.

ELIGIBILITY:
Inclusion Criteria:

* Case subject : at least one initial lateral ankle sprain more than 12 months before inclusion
* Case subject : at least one residual symptom among (1) giving way, (2) sensation of instability, (3) recurrent ankle sprain. This item is confirmed by a score inferior than 24 on the Chronic Ankle Instability Tool (CAIT)
* Case subject : Impact on activities of daily living and sport, confirmed by a score of less than 90% on the Foot and Ankle Ability Measure (FAAM) and less than 80% on FAAM-- - -- Control subject : matched by age and sex to case subjects

Exclusion Criteria:

* Surgery of one of the lower limbs less than 3 years ago
* Presence of heavy pain (EVA > 8) regardless of its origin
* Acute lateral ankle sprain less than 4 months before inclusion
* Neurological disorders of any kind
* Medical treatment (drugs) interfering with muscle tone, balance and proprioception disorders
* Pregnant or breastfeeding women
* Body mass index > 30
* Bilateral chronic ankle instability

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Adults (18-45 yrs) living in the northern part of France close to or in Lille, Saint-Omer and Amiens
Sampling Method: Non-Probability Sample
Enrollment: 4 (Actual)
Dates: Start 2019-10-24 (Actual); Primary Completion 2021-10-25 (Actual); Study Completion 2021-10-25 (Actual)

PRIMARY OUTCOMES:
Static balance tests | Baseline
  Static balance tests ( DLS and SLS (both ankles tested) ; Stabilometry) are composite measure
  * Centre of Pressure (COP) displacement (mm) ;
  * COP velocity (mm/s)
  * COP area (mm²)
  * COP time-to-boundary (TTB) (s)
  * Number of foot lifts (integer)
the Star Excursion Balance Test (SEBT) | Baseline
  Dynamic balance test : SEBT (both ankles tested) : are composite measure
  * Distance reached in anterior direction (% leg length)
  * Distance reached in posteromedial direction (% leg length)
  * Distance reached in posterolateral direction (% leg length)
  * Time used to reach (s)
  * COP displacement (mm)
  * COP velocity (s)
  * COP area (mm²)
  * COP time-to-boundary (TTB) (s)
Hop tests | Baseline
  Hop tests (both ankles tested) : SLHD et SH ; are composite measure
  * Distance reached (m)
  * Max inversion angle ankle joint (°)
  * Max internal rotation angle ankle joint (°)
  * Max vertical Ground Reaction Force (GRF) at landing (N)
  * Max lateral GRF (N)
  * Time used to complete 10 hops (s)
Strength tests (both ankles tested) | Baseline
  Isokinetic strength tests (both ankles tested) :
  * Plantar flexor peak torque (Nm)
  * Dorsiflexor peak torque (Nm)
  * Inversion peak torque (Nm)
  * Eversion Peak torque (Nm)

SECONDARY OUTCOMES:
Intra-class correlation coefficients (reproducibility test-retest) | Baseline and 1-4 weeks after baseline
  Intra-class correlation coefficients (reproducibility test-retest) calculated on the subset of the parameters identified by the main analysis.
  Recyclability of the functional clinical tests : Normality testing /Sample comparison

CONTACTS AND LOCATIONS:
Overall Officials: Alexandre Arnould, MD, Principal Investigator — University Hospital, Lille
Locations (1):
- CH Saint-Omer, institut audomarois de la chirurgie orthopédique et du sport, Saint-Omer, France